CLINICAL TRIAL: NCT01346501
Title: An Extended Observational Study (P12-707: HOPEFUL III Study) of Follow-up Survey (P12-069: HOPEFUL II Study) of the Study of Adalimumab (D2E7) for Prevention of Joint Destruction in Patients With Rheumatoid Arthritis in Japan (M06-859)
Brief Title: Special Investigation in Patients With Rheumatoid Arthritis (HOPEFUL III Study), a Follow-up Survey of Study P12-069
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-707
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Adalimumab: Participants with Rheumatoid Arthritis (RA) who continued adalimumab treatment after completion of study M06-859, participated in the observational period of studies P12-069 and P12-707.
  Other name for adalimumab is Humira.
- Non-adalimumab: Patients who discontinued adalimumab treatment after completion of the study M06-859.

SUMMARY:
The main objective of this study was to determine the ability to maintain response after discontinuation of adalimumab treatment and the secondary objective was to determine radiographic progression in participants participating in the study, including the percentage who displayed minimal progression.

DETAILED DESCRIPTION:
This was a two-arm, multi-center, Post Marketing Observational Study (PMOS) conducted in Japanese participants with Rheumatoid Arthritis (RA) who continued the one year observational period of study P12-069 (HOPEFUL II study; NCT01163292) and provided informed consent to participate in study P12-707 (HOPEFUL III study; NCT01346501), after completion of study M06-859 (HOPEFUL I study; NCT00870467). The study P12-707 provided an additional two years of observation for those participants who participated in study P12-069.

ELIGIBILITY:
Inclusion Criteria:

Participants with RA who continued the one year observational period of study P12-069 and provided informed consent to participate in study P12-707.

Exclusion Criteria:

Participants with RA who used biological agents other than adalimumab in the one year observational period of study P12-069.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Rheumatoid Arthritis (RA) who continued the one year observational period of study P12-069 and provided informed consent to participate in study P12-707.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2011-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Kurimoto, Study Director — AbbVie

REFERENCES:
- [Derived] Tanaka Y, Yamanaka H, Ishiguro N, Miyasaka N, Kawana K, Kimura J, Agata N, Takeuchi T. Low disease activity for up to 3 years after adalimumab discontinuation in patients with early rheumatoid arthritis: 2-year results of the HOPEFUL-3 Study. Arthritis Res Ther. 2017 Mar 14;19(1):56. doi: 10.1186/s13075-017-1264-6. PMID 28288682
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants with Rheumatoid Arthritis (RA) who continued adalimumab treatment after completion of study M06-859 (HOPEFUL I study; NCT00870467), participated in the observational period of studies P12-069 (HOPEFUL II study; NCT01163292) and P12-707 (HOPEFUL III study; NCT01346501).
- Non-adalimumab: Participants with RA who discontinued adalimumab treatment after completion of study M06-859, participated in the observational period of studies P12-069 and P12-707.
Period: Overall Study
Arm/Group | Adalimumab | Non-adalimumab
Started | 79 | 93
Completed | 68 | 80
Not Completed | 11 | 13
Not completed — Initiated Other Biological Agents | 3 | 1
Not completed — Other | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Adalimumab: Participants with RA who continued adalimumab treatment after completion of study M06-859, participated in the observational period of studies P12-069 and P12-707.
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Non-adalimumab | Total
Number analyzed (Participants) | 79 | 93 | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (13.6) | 55.2 (12.1) | 55.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 75 | 141
  Male | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Activity Score 28 - C-Reactive Protein (DAS28-CRP) Score < 3.2 After Discontinuation of Adalimumab Treatment
Description: The DAS28-CRP, a combined index that measured Rheumatoid Arthritis (RA) disease activity, was calculated based on the number of tender joint count (28 joints), the number of swollen joint count (28 joints), overall disease activity (using visual analog scale (VAS)), erythrocyte sedimentation rate (ESR), and C-Reactive protein (CRP). The DAS28-CRP scores ranged from 0 (no disease activity) to 9 (maximal disease activity); decrease in DAS28-CRP score indicated improvement of disease. In participants who discontinued treatment with adalimumab after sustained low disease activity (defined as DAS28-CRP score <3.2) in study M06-859, the percentage of participants who maintained DAS28-CRP score < 3.2 without disease flare (defined as DAS28-CRP score ≥ 3.2) during studies P12-069 and P12-707 was calculated.
Time Frame: At Week 0, Week 26, Week 52, Week 78, Week 104, Week 130, and Week 156
Population: The effectiveness analysis set was defined as all participants who had evaluable DAS28-CRP score during studies P12-069 and P12-707.
Measure: Number; unit: Percentage of participants
Groups:
- Non-adalimumab: Participants with RA who discontinued adalimumab treatment after completion of study M06-859 and sustained low disease activity (defined as DAS28-CRP score <3.2 at Week 46 and Week 52), participated in the observational period of studies P12-069 and P12-707.
Arm/Group | Non-adalimumab
Number analyzed (Participants) | 77
Percentage of participants
  Week 0 | 100.0
  Week 26 | 77.9
  Week 52 | 71.4
  Week 78 | 63.6
  Week 104 | 58.4
  Week 130 | 54.5
  Week 156 | 45.5

2. Primary Outcome: Percentage of Participants With Positive Serum Level of Matrix Metalloprotease-3 (MMP-3)
Description: MMP-3, a proteolytic enzyme that plays a pivotal role in joint destruction in RA was assessed during the study. MMP-3 serum level < 121 ng/mL in men and < 59.7 ng/mL in women was considered as the normal value. Data are presented as the percentage of participants with MMP-3 serum level greater than the normal value.
Time Frame: At Week 0, Week 26, Week 52, Week 78, Week 104, Week 130, Week 156, Week 182, and Week 208
Population: The effectiveness analysis set was defined as all participants who had evaluable MMP-3 score during studies P12-069 and P12-707.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab | Non-adalimumab
Number analyzed (Participants) | 77 | 84
Percentage of participants
  Week 0 | 79.2 | 67.9
  Week 26 (N=77, 83) | 53.2 | 38.6
  Week 52 | 37.7 | 27.4
  Week 78 (N=62, 57) | 38.7 | 36.8
  Week 104 (N=58, 66) | 19.0 | 42.4
  Week 130 (N=40, 46) | 25.0 | 32.6
  Week 156 (N=38, 52) | 28.9 | 32.7
  Week 182 (N=35, 38) | 20.0 | 23.7
  Week 208 (N=32, 43) | 18.8 | 30.2

3. Primary Outcome: Mean Health Assessment Questionnaire (HAQ) Score
Description: The HAQ score was a participant-reported questionnaire that measured quality of life in terms of physical function of participants with rheumatoid arthritis. It consisted of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past seven days using the following response categories (score): without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). The scores on each task were summed and averaged to provide an overall score from 0 to 3, where 0-1 represented mild disability and 2-3 represented severe disability. Data are presented as mean HAQ score +/- standard deviation with negative scores indicating improvement.
Time Frame: At Week 0, Week 26, Week 52, Week 78, Week 104, Week 130, Week 156, Week 182, and Week 208
Population: The effectiveness analysis set was defined as all participants who had evaluable HAQ score during studies P12-069 and P12-707.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab | Non-adalimumab
Number analyzed (Participants) | 72 | 83
Score on a scale
  Week 0 | 1.19 (0.70) | 1.04 (0.71)
  Week 26 (N=72, 82) | 0.48 (0.55) | 0.42 (0.46)
  Week 52 | 0.27 (0.35) | 0.25 (0.34)
  Week 78 (N=45, 48) | 0.13 (0.26) | 0.18 (0.32)
  Week 104 (N=55, 62) | 0.21 (0.30) | 0.23 (0.36)
  Week 130 (N=30, 44) | 0.18 (0.33) | 0.16 (0.27)
  Week 156 (N=28, 51) | 0.17 (0.35) | 0.30 (0.49)
  Week 182 (N=26, 33) | 0.20 (0.25) | 0.26 (0.43)
  Week 208 (N=24, 39) | 0.12 (0.33) | 0.19 (0.41)

4. Secondary Outcome: Percentage of Participants With Modified Total Sharp Score (mTSS) ≤ 0.5 and ≤ 1.5
Description: The mTSS, a method of assessing radiographs, was used to evaluate the level of joint destruction by disease. Digitized X-rays of hands and feet were obtained and scored on a scale ranging from 0 [no damage] to 5 [complete collapse or total destruction of joint] for erosion and 0 [no damage] to 4 [complete luxation of joint] for joint space narrowing. The scores on each task were summed and averaged to derive the total mTSS score ranging from 0 [normal] to 380 [maximal disease]. Large positive change in mTSS indicated disease progression; small positive/no change indicated slowing/halting of disease progression. The mTSS score ≤ 0.5 was defined as minimal radiographic progression. Data are presented as the percentage of the participants with mTSS ≤ 0.5 and ≤ 1.5 at the end of third year of the observation period (at Week 104 of P12-707).
Time Frame: 3 years
Population: The effectiveness analysis set was defined as all participants who had evaluable mTSS score during studies P12-069 and P12-707.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab | Non-adalimumab
Number analyzed (Participants) | 65 | 61
Percentage of participants
  mTSS ≤ 0.5 | 66.2 | 55.7
  mTSS ≤ 1.5 | 83.1 | 67.2

5. Secondary Outcome: Percentage of Participants With Adverse Drug Reactions and Serious Adverse Drug Reactions
Description: Adverse drug reactions (serious and non-serious) are adverse events for which the causal relationship between adalimumab and the event could not be ruled out. Adverse event was defined as any untoward or unintended medical occurrences (including abnormal laboratory findings), signs/symptoms, or diseases of the participant receiving adalimumab, regardless of causality of adalimumab treatment. Data are presented as percentage of participants.
Time Frame: From signing of informed consent until withdrawal of participant or starting a new biologic agent or up to approximately 2 years
Population: Safety was assessed in participants who received adalimumab in the observation period of studies P12-069 and P12-707, in routine clinical practice. Refer 'reporting group description' for the definition of safety analysis set.
Measure: Number; unit: Percentage of participants
Groups:
- Non-adalimumab: Participants with RA who discontinued adalimumab treatment after completion of study M06-859 and re-started adalimumab treatment during the observational period of studies P12-069 and P12-707.
Arm/Group | Adalimumab | Non-adalimumab
Number analyzed (Participants) | 79 | 22
Percentage of participants
  Adverse Drug Reactions | 16 | 2
  Serious Adverse Drug Reactions | 2 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent until withdrawal of participant or starting a new biologic agent or up to approximately 2 years
Description: The occurrence, type, severity, and relationship of adverse events to adalimumab were assessed. Safety was assessed in participants who received adalimumab in the observation period of studies P12-069 and P12-707, in routine clinical practice. Refer 'reporting group description' for the definition of safety analysis set.
Arm/Group | Adalimumab | Non-adalimumab
Serious Adverse Events (participants affected / at risk) | 3/79 | 1/22
Other Adverse Events (participants affected / at risk) | 25/79 | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=79) | Non-adalimumab (N=22)
Bronchiolitis (Infections and infestations) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=79) | Non-adalimumab (N=22)
Gastroenteritis viral (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 2 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Asthenopia (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.